CLINICAL TRIAL: NCT05448235
Title: the Effectiveness of the Thoracic Cage Mobilization on Chronic Obstructive Pulmonary Disease Patients
Brief Title: the Effectivness of the Thoracic Cage Mobilization on COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam omran Grase, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P. T. REC/012/003514
Record Dates: First submitted 2022-06-22; First posted 2022-07-07 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Thoracic cage mobilization; conventional treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: comparison between two groups one receive conventional treatment and other receives conventional treatment and thoracic mobilization
Who Masked: Participant, Outcomes Assessor
Masking Description: the patients , care provider and investigator do not know the groups receive treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment (Experimental): the patient will receive conventional treatment daily for up to one week
  Interventions: Other: conventional treatment
- thoracic cage mobilization (Experimental): the patient will receive thoracic cage mobilization added to conventional treatment daily for up to one week
  Interventions: Other: conventional treatment; Other: thoracic mobilization

INTERVENTIONS:
Other: conventional treatment — the patient will be asked to make pursed lip breathing (Breathe in for 2 seconds through his nose and Breathe out for 4 seconds through pursed lips)for 5-10 min ,3-4 times , 8-10 rep each cycle then asked to make diaphragmatic breathing exercise (Lie on his/her back and Inhale deeply through his/her nose for a count of three)for 5-10 min , 3-4 times , 8-10 repetition then postural drainage , furthermore the patient takes different position (prone to make percussion on lower lobes, side lying on anterior basal segment then sitting position on the upper lobe). After that a vibration on the chest (place a flat hand firmly atop the lung segment to be drained., and should apply light pressure and create a rapid, shaking movement) 1 min inhale and 5 time of repetition at the exhale and finally asked the patient to make productive cough for 5 times to get out the sputum.
Other: thoracic mobilization — we will use A SNAG to mobilization using type 3 oscillatory and sustain for 90 second, at first put the patient in 3 position (side lying to make mobilization of upper 6 ribs in downward direction then make on lower 6 ribs ,furthermore flexion of the thoracic and next rotation toward the midline then ask the patient to transfer to supine lying position and mobilize the sternum in downward direction the next mobilize the clavicle and ask the patient to take sitting position and put his hand on his head in adduction position and make extension on the thoracic vertebrae with inward mobilize with the investigator knees ,take each 4 vertebrae along the 12 thoracic vertebrae.
  Arms: thoracic cage mobilization

SUMMARY:
the study aims to investigate effectiveness of thoracic cage mobilizations on the chronic obstructive pulmonary diseases.

DETAILED DESCRIPTION:
COPD is a term for airflow restriction and growing shortness of breath caused by physiological deterioration. Elderly persons endure reduced respiratory function, stiffness in the joints and connective tissues of the rib cage, and increased thoracic Kyphosis as a result of COPD .breathlessness, cough, and sputum production are the most prevalent symptoms of COPD, while wheezing, chest tightness, and chest congestion are less common but nevertheless bothersome. The reported frequency, on the other hand, varies depending on the patient demographic and the severity of the disease. COPD is now the world's fourth greatest cause of mortality, but it is expected to rise to the third position by 2020.

Due to the obstruction and exhalation airflow is reduced, resulting in air trapping and hyperinflation. When the rate of minute ventilation or respiration is increased, for as during exercise, this becomes more apparent. Hyperinflation puts more strain on the respiratory muscles, forcing them to function in a restricted range of motion with a negative pressure/effort ratio, resulting in fatigue and increased shortness of breath. COPD patients avoid physical activity and adopt a more sedentary lifestyle than healthy older adults in order to prevent the distressing feeling of breathlessness. This, in turn, causes a vicious cycle of decreased exercise capacity, increased breathlessness during exercise, and more avoidance of exercise, and so on.

Active expiration, slow and deep breathing, pursed lips breathing, relaxation therapy, body positions such as forward leaning, inspiratory and expiratory muscle training, and diaphragmatic breathing are all examples of breathing techniques. Improvement of (regional) ventilation and gas exchange, decrease of dynamic hyperinflation, enhancement of respiratory muscle function, reduction of breathlessness, and improvement of exercise tolerance and quality of life are some of the goals of these procedures. Exercise capacity is impaired in COPD, both peak exercise capacity and functional exercise capacity. Besides lung hyperinflation and physical inactivity, ventilation-perfusion mismatch, hypoxemia, cardiovascular problems and muscular changes Reduced exercise capacity is a factor. One of the most important predictors of morbidity and mortality in COPD is functional exercise ability. and has a direct connection to everyday physical activities. Because rib cage mobility tends to be diminished with obstructive lung illness, PT appears to have a specific goal of rib cage joint mobility. Chest wall mobilization enhances chest wall mobility, lowers respiratory rate, raises tidal volume, improves ventilation gas exchange, reduces breathlessness, reduces work of breathing, and helps you relax. The rib cage mobilization is applied in three positions, supine ling, side lying and siding with arm abducted of the side to be mobilized.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease.
* Age >35 years.
* Received conventional medical treatment.
* the presence of at least two of the following three clinical criteria: a recent increase in breathlessness, sputum volume or sputum purulence.
* All enrolled patients either had previously been given a diagnosis of COPD by a physician or had at least a one-year history of chronic breathlessness or cough with sputum production

Exclusion Criteria:

* Admitted to the hospital, had been given a diagnosis of asthma or atrophy.
* Patients who had received oral or intravenous corticosteroid in the emergency department within the preceding 30 days.
* patient put on the mechanical ventilation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
ABG | up for one week
  to measure pH (7.35-7.45), PaO2 (75-100 mmHg), PaCO2 (35-45 mmHg), HCO3 (22-26 meq/L) and SaO2 (95-100%) we will measure these types of ABG Before and after the treatment and measure the difference before and after and compared it with the standard to detect the effect of the treatment on the lung function
chest expansion with tape measurement | up for one week
  using tape to measure chest exp ansion during inspiration and expiration at axillary level and at the level of T10 using CM units

SECONDARY OUTCOMES:
CAT questionnaire | up for one week
  to measure the patients status during treatment and after and It has eight categories (cough severity, presence of mucus, chest tightness, dyspnea, limits during domestic activities, social constraints, sleep, and energy restriction) with scores ranging from 0 (no impact) to 40 (significant impact) (severe impact) On a 7-point Likert scale (ranging from 1 to 7)
Dyspnea index | up for one week
  to measure the breathlessness after the treatment,used to determine levels of exertion and the Levels of shortness of breath (SOB): No SOB: can count to 15 (takes about 8 seconds) without taking a breath in the sequence.
  Mild SOB: can count to 15 but must take one short breath in the sequence. Moderate SOB; need to take 2 breaths to count to 15 in the sequence. Definite SOB: must take 3 breaths in the sequence of counting to 15. Severe SOB: unable to count

CONTACTS AND LOCATIONS:
Locations (1):
- Mariam omran Grase, Giza, Egypt